CLINICAL TRIAL: NCT04842045
Title: Recall of Experience and Conscious Awareness in Psilocybin Treatment of Depression (The RECAP Study): Pilot Phase in Healthy Adult Volunteers
Brief Title: Pilot RECAP Study in Healthy Volunteers
Acronym: RECAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0085; A532017 (Other: UW, Madison); SMPH/FAMILY MEDICINE (Other: UW, Madison); AAH3816 (Other: UWF- University of Wisconsin Foundation); PROTOCOL V7.0 10 OCT 2021 (Other: HS-IRB, UW Madison)
Record Dates: First submitted 2021-04-01; First posted 2021-04-12 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Psychedelic Experiences; Amnesia
Keywords: Memory; Amnesia; Healthy Volunteer
MeSH Terms: conditions — Amnesia | interventions — Psilocybin; Midazolam; Benzodiazepines

STUDY DESIGN:
Intervention Model Description: Open trial of a single 25 mg dose of psilocybin combined with repeated boluses of midazolam in medically and psychiatrically healthy volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Medically and psychiatrically healthy adults ages 21 to 65 years will receive a single 25 mg dose of psilocybin combined with repeated boluses of midazolam administered in a clinically supportive setting.
  Interventions: Drug: Psilocybin and Midazolam

INTERVENTIONS:
Drug: Psilocybin and Midazolam — The psilocybin used in this study is synthetically manufactured in a laboratory and meets quality specifications suitable for human research use. The active drug is encapsulated using a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of psilocybin.
  The midazolam in this study will be administered intravenously. The total dose administered to a given subject is dependent on the individual's level of amnesia, sedation scale score, age, and weight.
  Other Names: Psilocybine; Psilocibin; benzodiazepine

SUMMARY:
The primary objective of the RECAP Study Program is to investigate the role played by conscious experience in the antidepressant effects of the psychedelic agent psilocybin. This pilot dosing study (PILOT RECAP) is designed to determine the optimal dose of midazolam that allows a psychedelic experience to occur while inducing amnesia for the experience. This is an essential step required for subsequent evaluation of the role of memory for the psychedelic experience in the antidepressant effects of psilocybin in the full RECAP study.

DETAILED DESCRIPTION:
The PILOT RECAP Study will investigate the effect of co- administering the amnestic agent midazolam with a single 25 mg dose of psilocybin on the induction of a psychedelic experience and subsequent memory for the experience with the goal of identifying an optimal dosing regimen of midazolam that will allow a psychedelic experience to occur while also inducing amnesia for the experience. Identifying this midazolam dosing regimen will allow us in a subsequent stage of the RECAP program to test whether memory for the psychedelic experience is required/important for psilocybin to produce longer-term antidepressant effects. This is a phase 1 study in psychiatrically and medically healthy volunteers. Given this, there is no disease background for PILOT RECAP per se. However, the purpose of PILOT RECAP is to identify an optimal midazolam dosing schedule to be used in a subsequent study (RECAP) in patients with major depressive disorder (MDD).

The investigational treatment for PILOT RECAP is a single 25 mg dose of psilocybin combined with repeated intravenous (IV) boluses of midazolam dosed at levels known to maintain conscious experience while inducing subsequent amnesia for the experience upon its conclusion. Because PILOT RECAP is the first study to examine this drug combination, no data are currently available on this approach. Psilocybin + midazolam will be administered within a "Set and Setting" (SaS) protocol that provides psychoeducation and therapeutic support prior to, during, and following psychedelic dosing, and that has been standard procedure for recent studies of psilocybin in humans. It is believed that this SaS approach enhances clinical efficacy and safety. SaS is an integral component of the PILOT RECAP intervention.

The PILOT RECAP study will not enroll vulnerable populations. During this study, participants are asked to:

* Refrain from use of psychotropic medications. Use of such medications prior to psilocybin/midazolam dosing will result in a participant being discontinued from the study.
* Refrain from use of any illegal psychoactive substances from screening until study termination.
* Refrain from using legal psychoactive substance for the following defined time periods (the exception is caffeine):

  * Tobacco and Nicotine: from screening until study termination
  * Alcohol: 72 hours prior to the Dosing Visit

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 65 years at screening
* Medically healthy (does not meet criteria for an exclusionary medical condition)
* No current DSM-5 psychiatric diagnosis
* No current use of psychotropic medications
* Ability/willingness to complete all study activities
* Use of acceptable contraceptive methods (sexually active males and women of childbearing potential)
* Speaks and reads English
* No use of psychedelic drugs within prior 3 months of dosing visit
* Able to swallow oral medications

Exclusion Criteria:

* Pregnancy
* Current exclusionary medical illness
* Current DSM-5 psychiatric diagnosis and/or suicidal thoughts/behavior within prior 12 months
* Clinically significant safety lab abnormalities (i.e., Complete Blood Count with Differential, Comprehensive Metabolic Panel, and urinalysis)
* Clinically significant electrocardiogram (ECG)
* Hypertension or tachycardia
* First degree relative(s) with a history of schizophrenia, schizophreniform disorder, bipolar I disorder, bipolar II disorder, major depressive disorder with psychotic features

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Number of participants scoring >50 percent of normative scores on selected questions from the Altered States of Consciousness (ASC) questionnaire asked during the dosing session Day 0. | On Day 14
  Participants will complete a selection of several questions from the ASC questionnaire that strongly associate positively or negatively with later antidepressant effect of psilocybin in patients with treatment resistant depression or capture classic features of the psychedelic experience.
  During the dosing session, investigator will repeatedly ask selected items from the ASC scale to get a "real time" measure of what the participants are experiencing. Each of these items will be scored separately. Higher score are indicative of a more intense psychedelic experience.
Number of participants scoring < 50 percent on post-dosing Day 1 of the mean normative score of ASC data from healthy volunteers administered the ASC questionnaire post-dosing | On Day 15
  To assess the degree to which midazolam has induced amnesia for the psychedelic experience, participants will complete the full ASC.
  The ASC is a 94 item questionaire. In response to each item, participants are asked to mark their experience somewhere between 'No, not more than usual' to 'Yes, much more than usual'. Normal waking consciousness corresponds to a mark at the very left end of the scale, i.e. 'No, Not more than usual'.
  Responses marked more towards right side of the range are considered high on psychedelic experience.

SECONDARY OUTCOMES:
Accuracy on post-dosing Day 1 in recognizing ASC items asked during the dosing session Day 0 (number of correct versus distractor items) | On Day 15
  Participants will undergo a yes-no ASC recognition task regarding their memory for internally and externally focused phenomenological content of their experience.
Safety of psilocybin-midazolam co-administration assessed by number of adverse event incidences in each severity grade. | up to 4 weeks
  Adverse event grading will be done using Common Terminology Criteria for Adverse Event (CTCAE)Adverse events will be graded from Grade 1-5 depending on severity. Grade 1 - mild, grade 2 - moderate, grade 3 - severe, grade 4 - Life threatening, grade 5 - Fatal. Adverse events will be collected on an Adverse Event Log throughout the study.
Safety of psilocybin-midazolam co-administration assessed by number of participants requiring medical attention due to adverse events | up to 4 weeks
Safety of psilocybin-midazolam co-administration assessed by number of participants requiring psychiatric attention due to adverse events | up to 4 weeks
Safety of psilocybin-midazolam co-administration assessed by number of participants leading to withdrawal from study due to adverse events | up to 4 weeks
Safety of psilocybin-midazolam co-administration assessed by number of participants with severe adverse events | up to 4 weeks
Safety of psilocybin-midazolam co-administration assessed by number of participants with new concomitant medication due to adverse events | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Nicholas, MD,PHD, Principal Investigator — University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United State, 53715
Locations (1):
- UWHealth, 600 Highland Avenue, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No